CLINICAL TRIAL: NCT01381679
Title: Austrian Cholesterol Screening And Treatment II (ACT II)
Brief Title: Effect of Ezetimibe Treatment on Low-density Lipoprotein Cholesterol (LDL-C) Levels in Participants With Coronary Heart Disease (CHD) Already Treated With a Statin (MK-0653A-205 AM1)
Acronym: ACT II
Status: Completed | Type: Observational
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Other Study IDs: 0653A-205
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Results first posted 2012-03-22 (Estimated); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Ezetimibe

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All participants: Participants in whom LDL-C target levels have not been achieved and for whom ezetimibe therapy has been chosen.
  Interventions: Drug: Ezetimibe

INTERVENTIONS:
Drug: Ezetimibe — Ezetimibe was not mandatory and was prescribed as per routine prescription by physician.

SUMMARY:
This non-interventional longitudinal study is a follow-up of the Austrian Cholesterol Screening and Treatment project (ACT I), which assessed the cholesterol status, including achievement of the target levels applicable at that time (LDL levels <100 mg/dL), in participants with coronary heart disease (CHD) already being treated with a statin. In this study, participants without adequate LDL-cholesterol reduction with a statin underwent extension of therapy with ezetimibe with the goal of achieving target levels.

ELIGIBILITY:
Inclusion criteria:

* Participants in whom LDL-cholesterol target levels have not been achieved.
* Participants in whom a decision has been made by the physician to initiate treatment

with ezetimibe (longitudinal analyses). The treatment decision will be made prior to

and independent from inclusion of participants into this study.

- Participants with LDL cholesterol levels ≤113 mg/dl and a very high risk, which led to case-by-case approval of medication may be documented.

Exclusion criteria:

* Any condition which, in the opinion of the treating physician, precludes treatment with ezetimibe.
* In order not to interfere with data collection it is recommended not to include participants currently in a clinical trial.
* Previous and ongoing treatment with ezetimibe.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants without adequate LDL-cholesterol reduction with a statin, representative cross-section across all regions/parts of Austria (federal provinces, urban/rural areas, office-based internists/general practitioners)
Sampling Method: Non-Probability Sample
Enrollment: 1682 (Actual)
Dates: Start 2009-05; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

REFERENCES:
- [Derived] Pichler M, Lautsch D, Adler C, Bogl K, Drexel H, Eber B, Fauer C, Fochterle J, Foger B, Gansch K, Grafinger P, Lechleitner M, Ludvik B, Maurer G, Morz R, Paulweber B, Pfeiffer KP, Prager R, Stark G, Toplak H, Traindl O, Weitgasser R. Are there differences in LDL-C target value attainment in Austrian federal states? Yes! Wien Med Wochenschr. 2013 Dec;163(23-24):528-35. doi: 10.1007/s10354-013-0219-z. Epub 2013 Aug 27. PMID 23979353
- [Derived] Eber B, Lautsch D, Fauer C, Drexel H, Pfeiffer KP, Traindl O, Pichler M. Can LDL-cholesterol targets be achieved in a population at high risk? Results of the non-interventional study ACT II. Curr Med Res Opin. 2012 Sep;28(9):1447-54. doi: 10.1185/03007995.2012.717919. Epub 2012 Aug 16. PMID 22856551

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: Participants in whom low density lipoprotein cholesterol (LDL-C) target levels have not been achieved and for whom ezetimibe therapy has been chosen.
Period: Overall Study
Arm/Group | All Participants
Started | 1682
Completed | 794
Not Completed | 888
Not completed — Adverse Event | 3
Not completed — Lost to Follow-up | 885

BASELINE CHARACTERISTICS:
Arm/Group | All Participants
Number analyzed (Participants) | 1682
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.58 (10.4)
Sex/Gender, Customized [Number; unit: Participants]
  Males | 1003
  Females | 655
  Not Reported | 24
Region of Enrollment [Number; unit: participants]
  Austria | 1682

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving Individual LDL Cholesterol (LDL-C) Target Level
Description: Individual LDL-C target values were set according to the Austrian Cholesterol Consensus (ACC) 2007 for patients for patients suffering from coronary heart disease (CHD) or CHD equivalent in an office-based, routine medical care setting. Participants were categorized as either high-risk or very high-risk based on ACC criteria. The LDL-C target levels for each category were 100 mg/dL and 70 mg/dL, respectively
Time Frame: Up to 12 months
Measure: Number; unit: Participants
Arm/Group | All Participants
Number analyzed (Participants) | 1682
Participants | 678

2. Secondary Outcome: Change From Baseline in Total Cholesterol (TC) at Month 3
Time Frame: Baseline and Month 3
Population: Participants with baseline, follow-up visit 1 (3 months), and follow-up visit 2 (12 months) measurements for TC.
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | All Participants
Number analyzed (Participants) | 782
mg/dL | -46.6 (40.5) [-49.4 to -43.8]

3. Secondary Outcome: Change From Baseline in TC at Month 12
Time Frame: Baseline and Month 12
Population: Participants with baseline, follow-up visit 1 (3 months), and follow-up visit 2 (12 months) measurements for TC.
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | All Participants
Number analyzed (Participants) | 782
mg/dL | -54.5 (37.62) [-57.7 to -51.3]

4. Secondary Outcome: Change From Baseline in LDL-C at Month 3
Time Frame: Baseline and Month 3
Population: Participants with baseline, follow-up visit 1 (3 months), and follow-up visit 2 (12 months) measurements for LDL-C.
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | All Participants
Number analyzed (Participants) | 750
mg/dL | -41.7 (31.81) [-44.2 to -39.3]

5. Secondary Outcome: Change From Baseline in LDL-C at Month 12
Time Frame: Baseline and Month 12
Population: Participants with baseline, follow-up visit 1 (3 months), and follow-up visit 2 (12 months) measurements for LDL-C.
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | All Participants
Number analyzed (Participants) | 750
mg/dL | -49.3 (26.64) [-51.9 to -46.7]

6. Secondary Outcome: Change From Baseline in High-density Lipoprotein Cholesterol (HDL-C) at Month 3
Time Frame: Baseline and Month 3
Population: Participants with baseline, follow-up visit 1 (3 months), and follow-up visit 2 (12 months) measurements for HDL-C.
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | All Participants
Number analyzed (Participants) | 774
mg/dL | 2.8 (14.17) [2.0 to 3.6]

7. Secondary Outcome: Change From Baseline in HDL-C at Month 12
Time Frame: Baseline and Month 12
Population: Participants with baseline, follow-up visit 1 (3 months), and follow-up visit 2 (12 months) measurements for HDL-C.
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | All Participants
Number analyzed (Participants) | 774
mg/dL | 4.0 (15.05) [3.1 to 5.0]

8. Secondary Outcome: Change From Baseline in Triglycerides (TG) at Month 3
Time Frame: Baseline and Month 3
Population: Participants with baseline, follow-up visit 1 (3 months), and follow-up visit 2 (12 months) measurements for TG.
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | All Participants
Number analyzed (Participants) | 756
mg/dL | -33.8 (82.51) [-41.1 to -26.6]

9. Secondary Outcome: Change From Baseline in TG at Month 12
Time Frame: Baseline and Month 12
Population: Participants with baseline, follow-up visit 1 (3 months), and follow-up visit 2 (12 months) measurements for TG.
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | All Participants
Number analyzed (Participants) | 756
mg/dL | -43.9 (75.06) [-51.5 to -36.4]

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | All Participants
Serious Adverse Events (participants affected / at risk) | 3/1682
Other Adverse Events (participants affected / at risk) | 0/1682
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Participants (N=1682)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bronchial Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less